CLINICAL TRIAL: NCT04337905
Title: A New Development Diagnostic Tool for ADHD: A VR Approach
Brief Title: Virtual Reality (VR) Diagnostic Tool for Attention Deficits/Hyperactivity Disorder (ADHD)
Acronym: New
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tjhin Wiguna (Other)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other); Dr Cipto Mangunkusumo General Hospital (Other); Binus University International (Unknown)
Responsible Party: Sponsor-Investigator, Tjhin Wiguna, Prof. Dr. dr., Dr Cipto Mangunkusumo General Hospital
Organization: Dr Cipto Mangunkusumo General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ADHD-VR
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: ADHD; Executive Dysfunction
Keywords: ADHD; virtual reality,; diagnostic tool; neuropsychological test; Indonesia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: There is two group of children:
  1. Group 1: Children with ADHD
  2. Group 2: Children without ADHD as a control group
  Both group will running the ADHD-VR diagnostic test and goes to diagnosis by child psychiatrist. The outcomes that were analyzed:
  1. The sensitivity, specificity and Likelihood ratio of the ADHD-VR diagnostic test in detecting the ADHD clinical symptoms and executive function
  2. Content validity of the ADHD-VR diagnostic test
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator blind to the ADHD-VR diagnostic test results The care provider blind to the ADHD-VR diagnostic test results The ADHD-VR assessor blind to the ADHD diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with ADHD (Experimental): Children with ADHD that running the ADHD-VR diagnostic test and also did the psychiatric examination to determine the ADHD diagnosis and to rule out other mental disorders
  Interventions: Device: ADHD-VR diagnosis tool
- Children without ADHD (Active Comparator): Healthy children that also running the ADHD-VR diagnostic test and also psyhchiatric examination to rule out the ADHD diagnosis and other mental disorders
  Interventions: Device: ADHD-VR diagnosis tool

INTERVENTIONS:
Device: ADHD-VR diagnosis tool — Since that time and in accordance with the application area, several definitions have been formulated: for example, Fuchs and Bishop (1992) defined VR as "real-time interactive graphics with 3D models, combined with a display technology that gives the user the immersion in the model world and direct manipulation"; Gigante (1993) described VR as "The illusion of participation in a synthetic environment rather than external observation of such an environment. VR relies on a 3D, stereoscopic head-tracker displays, hand/body tracking and binaural sound. VR is an immersive, multi-sensory experience"; and "Virtual reality refers to immersive, interactive, multi-sensory, viewer-centered, 3D computer generated environments and the combination of technologies required building environments".

SUMMARY:
Attention deficit/ hyperactivity disorder (ADHD) is a common neurodevelopmental disorder. The common diagnostic of ADHD is based on psychiatric examination and interview. So far, there is not any other diagnostic tool for ADHD nowadays. Therefore, virtual reality (VR) technology can be used as a stimulus, replacing real stimuli, recreating experiences, which are in the real world would be impossible. Consequently, ADHD-VR diagnostic tool development should be started to justify the ADHD diagnosis in psychiatric out-patient clinical services.

DETAILED DESCRIPTION:
Diagnostic test is a very essential in modern medical practices, especially in child and adolescent psychiatry field because the main diagnostic tool is only based on psychiatry interview and observation. Using Diagnostic tool can help a confirmation towards specific clinical diagnosis, provide more evidence for eliminating one diagnosis versus another, provide more evidence for parents, or to rule out the differential diagnosis. Even though psychiatric examination is the main approach on ADHD diagnostic procedure, however the laboratory testing or imaging examination is also used especially to rule out the general medical condition or to find out any medical conditions that mimic ADHD but not to facilitate the ADHD diagnosis per se. Nowadays, the expand study in biological psychiatry has found a lot of biological markers in ADHD as well; but none is really sensitive and specific for ADHD diagnostic test. Therefore, there should be another approach for developing diagnostic tool in ADHD. VR is one of the best approach bacasue these days, because VR as an ADHD diagnostic tool could create and replace real stimuli, recreating experiences, which could not be observed by the clinician at the out-patient clinic.

ELIGIBILITY:
Inclusion Criteria for ADHD group:

* Children with ADHD drug naive
* Parent willing to participate in the study by signing informed consent
* Children willing to participate the ADHD-VR diagnostic tool for at least 30 minutes

Exclusion Criteria:

* Having untreated chronic physical illnesses
* Having other mental disorders except ADHD

Inclusion Criteria for healthy children group:

* Do not have any mental disorder
* Do not have untreated chronic physical illnesses
* Parent willing to participate in the study by signing informed consent
* Children willing to participate the ADHD-VR diagnostic tool for at least 30 minutes

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-05-25 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of ADHD-VR diagnostic tool towards ADHD clinical symptoms | up to 30 minutes
  The comparing between the ADHD-VR diagnostic test results and expert judgement on ADHD diagnosis
The sensitivity and specificity of ADHD-VR diagnostic tool towards executive function | up to 30 minues
  Comparing between the ADHD-VR diagnostic test results and Behavior Rating Inventory for Executive Function Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tjhin Wiguna, PhD, Principal Investigator — Dr Cipto Mangunkusumo General Hospital
Locations (1):
- dr. Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
No decided yet